CLINICAL TRIAL: NCT05557461
Title: Assessment of Fluid Responsiveness in Septic Shock Patients, Can End-tidal co2 Measurement Help?, a Prospective Observational Study
Brief Title: Assessment of Fluid Responsiveness in Septic Shock Patients, Can End-tidal co2 Measurement Help?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, hüseyin özkarakaş, intensive care specialist Medical Doctor, Bozyaka Training and Research Hospital
Other Study IDs: huseyinetco2
Record Dates: First submitted 2022-08-19; First posted 2022-09-28 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Septic Shock; Hypovolemia; Sepsis
Keywords: passive leg raise; capnography; fluid therapy; echocardiography; Fluid Responsiveness
MeSH Terms: conditions — Shock, Septic; Hypovolemia; Sepsis | interventions — Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group-1: group with fluid responsiveness in passive leg raise test After the patients are in a semi-sitting position (at least 2 minutes), two healthcare professionals will take the supine position and then lift their legs 45 degrees, wait for 2 minutes and return to the initial position.
  10% change in stroke volume will be considered positive and patients will be divided into 2 groups as fluid-responsive and non-responsive.
  Interventions: Device: End-tifdal co2, systolic, diastolic blood pressure, ppv values and vci distensibility
- Group-2: group with no fluid response in passive leg raise test After the patients are in a semi-sitting position (at least 2 minutes), two healthcare professionals will take the supine position and then lift their legs 45 degrees, wait for 2 minutes and return to the initial position.
  10% change in stroke volume will be considered positive and patients will be divided into 2 groups as fluid-responsive and non-responsive.
  Interventions: Device: End-tifdal co2, systolic, diastolic blood pressure, ppv values and vci distensibility

INTERVENTIONS:
Device: End-tifdal co2, systolic, diastolic blood pressure, ppv values and vci distensibility — (0,1,3,5 minutes measurements will be taken) measured before and after the test will be recorded and compared.
  Cardiac output and stroke volume variation, vci distensibility will be measured and recorded by a specialist cardiologist using siemens ocuson cv70 (Siemens AG Medical Solutions, Henkestrasse, the Germany) echocardiography before and after the test.

SUMMARY:
Fluid therapy is important in patients with sepsis and septic shock. There are many invasive and non-invasive methods to assess fluid responsiveness in patients. The specificities and sensitivities of these methods are highly variable. The reason for our study was to determine end-tidal co2 and fluid responsiveness in septic shock patients. The aim of the study was to evaluate the fluid response using the End-tidal CO2 difference in septic shock patients receiving intubated mechanical ventilation support.

DETAILED DESCRIPTION:
End-tidal CO2 is a parameter that can be easily measured with our non-invasively available monitors. If results are positive, fluid response of patients can be measured with a non-invasive, easy-to-apply method.

The significance of end-tidal CO2 will be confirmed by the passive leg raise test. Assessment of fluid responsiveness with the passive leg raise test is currently seen as the non-invasive reference test used.

It has proven its accuracy and reliability in many studies. In the passive leg raise test, end-tidal CO2 will be compared between the group with and without fluid responsiveness.

Scope of the study: Patients hospitalized in the general and reanimation intensive care units of our hospital and diagnosed with septic shock for any reason.

Method(s) to be applied: All patients diagnosed with septic shock will be included in the study.

The passive leg raise test, will be applied to the patients, and cardiac output and end-tidal CO2 changes will be recorded with transthoracic echocardiography before and after.

Fluid responsiveness is considered to be present in patients whose stroke volume variation output change measured by echocardiography increases by 10% or more after the passive leg raise test.

Patients will be divided into 2 groups according to fluid responsiveness. Group-1 group with fluid responsiveness in passive leg raise test, Group-2 group with no fluid response in passive leg raise test. End-tidal CO2 will be compared between groups.

Passive leg raise test: After the patients are in a semi-sitting position (at least 2 minutes), two healthcare professionals will take the supine position and then lift their legs 45 degrees, wait for 2 minutes and return to the initial position.

With this maneuver, it is anticipated that approximately 150-300 ml of autotransfusion will be administered to the patient.

Statistical analyzes will be made with the SPSS 21 program. Normally distributed data will be expressed as mean ± standard deviation, non-normally distributed data will be expressed as median. Categorical data will be expressed as a percentage. The difference between the mean and median values will be evaluated according to the distribution of the data by Student's t or Mann-Whitney U test. Categorical data will be evaluated with the chi-square test. A p value <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* in circulatory shock
* Hemodynamically stable for 10 minutes (whether or not he takes vasoactive drugs)
* Followed in mechanical ventilation with invasive arterial monitoring

Exclusion Criteria:

* pregnant
* Heart cannot be visualized by echocardiography
* Patients for whom passive leg raise test cannot be performed
* Bilateral lower extremity amputation
* Patients who are hemodynamically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the general and reanimation intensive care units of our hospital and diagnosed with septic shock for any reason
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-02-27 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
end tidal co2 | Recording will be made immediately before the passive leg raise test.
  the level of carbon dioxide that is released at the end of an exhaled breath
end tidal co2 | Recording will be made at the 1st minute after the end of the test.
  the level of carbon dioxide that is released at the end of an exhaled breath
end tidal co2 | Recording will be made 3rd minute after the end of the test.
  the level of carbon dioxide that is released at the end of an exhaled breath

SECONDARY OUTCOMES:
diastolic blood pressure | Recording will be made immediately before the passive leg raise test.
diastolic blood pressure | Recording will be made at the 1st minute after the end of the test.
diastolic blood pressure | Recording will be made 3rd minute after the end of the test.
systolic blood pressure | Recording will be made immediately before the passive leg raise test.
systolic blood pressure | Recording will be made at the 1st minute after the end of the test.
systolic blood pressure | Recording will be made 3rd minute after the end of the test.
ppv values | Recording will be made immediately before the passive leg raise test.
  Pulse pressure variation
ppv values | Recording will be made at the 1st minute after the end of the test.
  Pulse pressure variation
ppv values | Recording will be made 3rd minute after the end of the test.
  Pulse pressure variation
vci distensibility | Recording will be made immediately before the passive leg raise test.
  Distensibility Index of Inferior Vena Cava
vci distensibility | Recording will be made at the 1st minute after the end of the test.
  Distensibility Index of Inferior Vena Cava
vci distensibility | Recording will be made 3rd minute after the end of the test.
  Distensibility Index of Inferior Vena Cava

CONTACTS AND LOCATIONS:
Overall Officials: Zeki T Tekgül, Assoc Prof, Study Chair — Izmir Bozyaka Training and Research Hospital; Özkan özmuk, MD, Study Chair — Izmir Bozyaka Training and Research Hospital; Çağrı Yeşilnacar, MD, Study Chair — Izmir Bozyaka Training and Research Hospital; Oğuz Uçar, MD, Study Chair — Izmir Bozyaka Training and Research Hospital; Mehmet Uğur Bilgin, MD, Study Chair — Izmir Bozyaka Training and Research Hospital
Locations (1):
- UHS Izmir Bozyaka Education and Research Hospital, Izmir, Karabağlar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monnet X, Marik P, Teboul JL. Passive leg raising for predicting fluid responsiveness: a systematic review and meta-analysis. Intensive Care Med. 2016 Dec;42(12):1935-1947. doi: 10.1007/s00134-015-4134-1. Epub 2016 Jan 29. PMID 26825952
- [Background] Arango-Granados MC, Zarama Cordoba V, Castro Llanos AM, Bustamante Cristancho LA. Evaluation of end-tidal carbon dioxide gradient as a predictor of volume responsiveness in spontaneously breathing healthy adults. Intensive Care Med Exp. 2018 Jul 30;6(1):21. doi: 10.1186/s40635-018-0187-0. PMID 30062599
- [Background] Toupin F, Clairoux A, Deschamps A, Lebon JS, Lamarche Y, Lambert J, Fortier A, Denault AY. Assessment of fluid responsiveness with end-tidal carbon dioxide using a simplified passive leg raising maneuver: a prospective observational study. Can J Anaesth. 2016 Sep;63(9):1033-41. doi: 10.1007/s12630-016-0677-z. Epub 2016 Jun 15. PMID 27307176